CLINICAL TRIAL: NCT07220577
Title: A Multicenter, Randomized, Participant- and Investigator -Blinded, Placebo-controlled, Phase 2a Study to Assess the Efficacy, Safety and Tolerability of GIA632 in Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: Phase 2a Study to Assess the Efficacy,Safety and Tolerability of GIA632 in Adult Participants With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGIA632A12201; 2025-521503-43 (Other: EU CTIS)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: Phase 2; interventional; atopic dermatitis; efficacy; safety
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GIA632 (Experimental): Active treatment arm
  Interventions: Drug: GIA632
- Placebo (Placebo Comparator): Placebo treatment arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GIA632 — Active treatment arm
  Arms: GIA632
Other: Placebo — Placebo treatment arm
  Arms: Placebo

SUMMARY:
The main purpose of this Ph2a study is to evaluate the preliminary efficacy, safety and tolerability of GIA632 when administered to adult participants with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel-group, non-confirmatory, investigator and participant blinded study in adult participants with moderate to severe AD.

ELIGIBILITY:
Key Inclusion Criteria:

* Able and willing to sign the informed consent form
* Patients with a diagnosis of atopic dermatitis and disease for at least 1 year
* Moderate to severe atopic dermatitis

Key Exclusion Criteria:

* Participants with a clinically significant medical condition or infectious disease (as specified in the protocol)
* Participants with any clinically significant abnormal clinical laboratory tests, vital signs, physical examination or ECG
* Participant with any other active inflammatory skin disease would interfere with the appropriate assessment of atopic dermatitis in the opinion of the investigator
* Participants with any chronic, uncontrolled medical condition, which would put the participant at increased risk during the study (e.g., uncontrolled: diabetes, hypertension)
* Participants with any clinically unstable disease states that would likely require systemic corticosteroids (e.g., uncontrolled asthma)
* Women of childbearing potential unless they are using highly effective methods of contraception (failure rate < 1% per year) while taking study treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2027-09-13 (Estimated)

PRIMARY OUTCOMES:
IGA response at Week 16 defined as clear (0) or almost clear (1) score with at least a 2 point-reduction from baseline | Baseline, Week 16
  To assess the efficacy of GIA632 compared to placebo at week 16

CONTACTS AND LOCATIONS:
Locations (15):
- United States (3):
  - Ctr for Dermatology Clinical Res, Fremont, California
  - Aesthetics Skin Care Dermatologic Surgery, Rockville, Maryland
  - Care Access Hoboken, Hoboken, New Jersey
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Dijon, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Malaysia (3):
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Gdansk, Poland
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.